CLINICAL TRIAL: NCT07235969
Title: A Single-center, Randomized, Parallel-group Study to Compare the Efficacy of Psychologically Informed Physical Therapy, Tendon-Specific Exercise Program and Routine Physical Therapy in Prolonged Unilateral Shoulder Pain: RESSPECT Study
Brief Title: New Therapeutic Interventions and Imaging Techniques for Prolonged Shoulder Disorders
Acronym: RESSPECT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 151/2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Shoulder Pain; Pain Management; Physical Therapy
Keywords: Pain Management; Psychologically Informed Physical Therapy; Magnetic resonance fingerprinting; Diagnostic Imaging; Microvascular Flow Imaging; Tendon-Specific Exercise Program; Shear Wave Elastography
MeSH Terms: conditions — Shoulder Pain; Agnosia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The participants are not masked to their respective treatment, but are masked to the treatment other study groups receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Occupational physiotherapy (control group) (Active Comparator)
  Interventions: Other: Occupational health care led physiotherapy
- Physiotherapist-guided Tendon-Specific Exercise Program (TSEP) (Experimental)
  Interventions: Other: Tendon-Specific Exercise Program (TSEP)
- Physiotherapist-guided Psychologically Informed Physical Therapy (PIPT) (Experimental)
  Interventions: Other: Psychologically Informed Physical Therapy (PIPT)

INTERVENTIONS:
Other: Tendon-Specific Exercise Program (TSEP) — The aims of the TSEP are to improve RC muscle strength and increase tendon stiffness. The principles of exercise intervention are based on High-Loading Tendon Exercise (HLTE) and Heavy Slow Resistance (HSR) Training programs, and the Pain Monitoring Model (PMM).
  Arms: Physiotherapist-guided Tendon-Specific Exercise Program (TSEP)
Other: Psychologically Informed Physical Therapy (PIPT) — The aims of PIPT are biopsychosocial framework, patient-centered care and communication, good patient-therapist relationship, and consideration of patient's beliefs, fears and attitudes, behavior change, and guided self-management.
  Arms: Physiotherapist-guided Psychologically Informed Physical Therapy (PIPT)
Other: Occupational health care led physiotherapy — Subjects will be advised to contact the occupational health care to receive routine physiotherapy for their shoulder symptoms.
  Arms: Occupational physiotherapy (control group)

SUMMARY:
The RESSPECT study compares three types of physical therapy for adults aged 20-60 years with prolonged shoulder disorders, aiming to find better ways to help people recover and improve daily function. The study also examines modern imaging tests (X-ray, ultrasound, MRI) to see how well imaging findings match real symptoms, and tests new imaging technologies that may provide a more accurate diagnosis. The study improves future shoulder pain care by addressing both physical and psychological factors and advancing diagnostic imaging.

Participants are randomly assigned to one of three groups:

1. Routine physical therapy (usual occupational care),
2. Tendon-Specific Exercise Program (TSEP): targeted exercises to build shoulder strength and
3. Psychologically Informed Physical Therapy (PIPT): combining physical rehabilitation with advice and emotional support.

All participants get complete imaging of both shoulders and a clinical evaluation by a physiotherapist at the start of the study. Complete imaging is also done for all participants after twelve months. Surveys about pain, movement, mood, sleep, and quality of life are collected electronically at the start of the study, and at three, six, twelve, and 36 months. The main outcome is how well each person resumes everyday activities affected by shoulder pain (Patient-Specific Functional Scale, PSFS).

Group 1 will receive routine occupationally led physiotherapy, and groups 2 and 3 will receive five physiotherapist-guided sessions during the first six month-period. Advanced imaging techniques will deployed in conjunction with standard imaging methods and compared to see whether new technologies help explain symptoms or guide care.

To join, participants must have had prolonged shoulder disorders in one shoulder for at least four consecutive weeks, be employed or self-employed, and be willing to take part in rehabilitation activities. Certain medical conditions, prior surgery, and pregnancy are exclusion criteria. Inclusion and exclusion criteria are systematically reviewed in a structured phone interview at the start of the study. Baseline imaging is also viewed preliminarily for certain conditions which would require urgent medical care. If necessary, participants are contacted, informed and subsequently excluded from the study.

The trial takes place at Oulu University Hospital, Finland. Approximately 300 people are recruited to the study via local ads. Informed consent is required for the study, and participants can withdraw at any time. All procedures meet ethical standards.

This study will help determine:

1. Which therapy works best overall
2. Whether some people benefit more from certain therapies
3. If imaging findings help predict outcomes or aid treatment decisions
4. Whether new imaging technology improves diagnosis

DETAILED DESCRIPTION:
Shoulder complaints are one of the most common musculoskeletal ailments in general practice and a leading cause of work absence. While imaging findings are common in both symptomatic and asymptomatic shoulders, patient-specific characteristics such as obesity, depression and physical labor are risk factors for reported shoulder symptoms. Usually, general exercises have been considered useful in treating patients with shoulder symptoms, with the lack of evidence of specific tendon exercises. Biopsychosocial model is recommended in treatment of disabling musculoskeletal pain and to enhance self-management. Psychologically Informed Physical Therapy (PIPT) considers biopsychosocial framework in patient management, but it has not extensively been studied among patients with shoulder symptoms.

The RESSPECT study is a single-center randomized longitudinal parallel-group superiority study that aims to evaluate the effectiveness and cost-effectiveness of routine and specific physical therapy interventions, focusing on tendon and biopsychosocial rehabilitation. In total, 300 study participants will be recruited from the North Ostrobothnia region through local advertisements. The initial eligibility assessment will be done using a structured telephone interview, where potential participants will be evaluated against the inclusion and exclusion criteria, and the written information of the study will be distributed. The study includes diagnostic imaging at baseline and at 12 months, a baseline clinical PT visit for all participants and either routine occupationally led PT or five PT-guided sessions for the two interventional groups during the first six month-period, in three similar-sized groups. Electronic surveys will be asked to be filled at baseline prior to clinical visit as well as at three, six, twelve- and 36-months follow-up time points. Before the clinical visit, baseline imaging and patient records are preliminarily reviewed for exclusion criteria and, where applicable, participants are contacted and removed from the study.

The surveys cover a wide range of questions related to general health, details of employment, illnesses and medications, shoulder as well as generalized pain, demographic and socioeconomic factors, lifestyle, fear of pain and functional capacity. The electronic surveys also include validated Finnish versions of several structured questionnaires. Surveys are filled in and study data will be collected using an electronic data collection system (REDCap). In the baseline survey, participants are also instructed to fill in a traditional pain drawing. Follow-up surveys have additional questions regarding trauma, upper limb fractures and dislocations and newly diagnosed illnesses as well as their respective potentially caused shoulder dysfunction, planned or performed procedures of the upper limb and their nature, and confirmed or possible pregnancy. The personal participant-named activities in the PSFS will be carried over from the baseline questionnaire to the follow-up surveys, and the PSFS acts as the primary outcome of the study. As an active occupational health care service is required for study enrollment, follow-up surveys also ask participants to check and report their prior PT, physician and other healthcare professional visits regarding shoulder symptoms as well as prior shoulder imaging from their respective occupational health care mobile applications, which are widely available in the Finnish occupational health care system.

Bilateral shoulder imaging using conventional radiographs (CRs), multiparametric US and contrast-enhanced MRI will be conducted for inter-modality comparison as well as correlative studies between imaging findings, symptoms and effectiveness of different rehabilitation interventions. The added diagnostic capability of modern US and MRI technological advances will also be tested, focusing on RC structures, against conventional US and MRI. Bilateral shoulder CRs will be imaged in three projections. From the CRs, shoulder anatomy, glenohumeral and acromioclavicular degeneration, indirect signs of RC tears as well as potential calcium deposits will be evaluated. Osteoarthritis of the glenohumeral joint will be graded according to Kellgren-Lawrence classification (grades 0 to 4), and osteoarthritis of the acromioclavicular joint will be graded according to Petersson classification (grades 0-3). Bilateral static and dynamic shoulder US will be imaged using high-end US machines with high frequency linear probes by highly experienced sonographers with at least 10 years of experience in musculoskeletal US. US will be done following the musculoskeletal US technical guidelines published by the European Society of Musculoskeletal Radiology, and shear wave elastography and superb microvascular imaging techniques will be implemented during the US examination. Bilateral contrast-enhanced shoulder MRI will be imaged using a 3T scanner and a dedicated shoulder coil. Non-contrast MRI sequences including Magnetic Resonance Fingerprinting will be imaged first for both shoulders, after which contrast enhanced sequences will be imaged in succession, starting with the symptomatic shoulder.

The number of individuals assessed for eligibility will be recorded and reported in published results. The projected progress of all enrolled participants will be scheduled at the time of recruitment to ensure the timely preliminary evaluation of imaging studies, rehabilitation and electronic surveys. The preliminary review of participant imaging, electronic surveys and patient records will be done by the primary investigator, a musculoskeletal radiology fellow, with available consultation from a board-certified musculoskeletal radiologist with eleven of years of experience and a physiatrist with ten years of experience. Considering the biopsychosocial concept of pain, information about imaging findings is not given to the participants during the study, however, participants are ensured that they are informed of all imaging findings requiring urgent medical attention, followed by exclusion from the study if applicable. This information is separately highlighted in the consent form. Participant retention will be improved and drop-out reduced by electronic reminders of surveys, PT sessions and the 12-month imaging. Every reasonable effort to schedule sessions at participant-compatible times will be made and possibilities for rescheduling will be offered. In case of no-show, a request to schedule a new appointment will be sent.

ELIGIBILITY:
Inclusion Criteria:

* Age of 20-60 years
* Active participation in the workforce (employed or entrepreneur)
* Active occupational health care services available
* Daily unilateral shoulder pain for at least four consecutive weeks
* Willingness to participate in independent rehabilitation and PT visits

Exclusion Criteria:

* Bilateral shoulder pain
* Previous humerus fracture or current acute upper limb injury
* Prolonged dysfunction or pain of the upper limb attributable to trauma, neurologic disease or cervical spine disorders
* Diagnosed musculoskeletal disorders affecting the upper limb (e.g. rheumatoid arthritis)
* Severe disability, mental or memory disorder
* Advanced cancer
* History of shoulder PT or corticosteroid injection in the last six months
* Previous or planned shoulder surgery
* Confirmed or possible pregnancy
* Contraindications to MRI
* Severe chronic kidney disease
* Evidence unaccounted malignancy or other exclusionary findings in the initial eligibility assessment on either side

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Patient-Specific Functional Scale | From baseline to the end of the follow-up at 36 months
  The personal participant-named activities in the structured PSFS form at baseline will be carried over to the follow-up surveys, against which patients will do the scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Antti Kemppainen, Dr., Principal Investigator — University of Oulu
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in a publication, upon reasonable request and in compliance with EU's GDPR and Finland's Secondary Use Act
Supporting Information: Study Protocol
Time Frame: Beginning after the publication of results and ending 3 years after.